CLINICAL TRIAL: NCT03927157
Title: A Regional, Multicentre, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Adults With Severe Uncontrolled Asthma
Brief Title: Study to Evaluate Tezepelumab in Adults With Severe Uncontrolled Asthma
Acronym: DIRECTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00021
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Asthma; Uncontrolled Asthma; Severe Uncontrolled Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either tezepelumab or matching placebo both administered subcutaneously.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab: Tezepelumab subcutaneous injection
  Interventions: Biological: Experimental: Tezepelumab
- Placebo (Placebo Comparator): Placebo: Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Experimental: Tezepelumab — Tezepelumab subcutaneous injection
  Other Names: Tezepelumab
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A Regional, Multicentre, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Adults with Severe Uncontrolled Asthma

DETAILED DESCRIPTION:
This is a regional, multicentre, randomized, double-blind, placebo controlled, parallel group, phase 3 study designed to evaluate the efficacy and safety of 210 mg Q4W (SC) of tezepelumab in adults with severe, uncontrolled asthma on medium to high-dose ICS and at least one additional asthma controller medication with or without OCS. Approximately 396 participants will be randomized regionally (China/non-China). Participants will receive tezepelumab, or placebo, administered via subcutaneous injection at the study site, over a 52-week treatment period. The study also includes a post-treatment follow-up period of 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age. 18-80
* Documented physician-diagnosed asthma for at least 12 months
* Participants who have received a physician-prescribed asthma controller medication with medium or high dose ICS for at least 6 months.
* Documented treatment with a total daily dose of either medium or high dose ICS (≥ 500 µg fluticasone propionate dry powder formulation equivalent total daily dose) for at least 3 months.
* At least one additional maintenance asthma controller medication is required according to standard practice of care and must be documented for at least 3 months.
* Morning pre-BD FEV1 <80% predicted normal
* Evidence of asthma as documented by either: Documented historical reversibility of FEV1 ≥12% and ≥200 mL in the previous 12 months OR Post-BD (albuterol/salbutamol) reversibility of FEV1 ≥12% and ≥200 mL during screening.
* Documented history of at least 2 asthma exacerbation events within 12 months, and at least one of the exacerbations should occur during the treatment of medium-to-high dose ICS.
* ACQ-6 score ≥1.5 at screening and on day of randomization

Exclusion Criteria:

* Pulmonary disease other than asthma.
* History of cancer.
* History of a clinically significant infection.
* Current smokers or participants with smoking history ≥10 pack-yrs.
* History of chronic alcohol or drug abuse within 12 months.
* Hepatitis B, C or HIV.
* Pregnant or breastfeeding.
* History of anaphylaxis following any biologic therapy.
* participant randomized in the current study or previous tezepelumab studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, Bachelor, Principal Investigator — Guangzhou institute of Respiratory Disease, China
Locations (50):
- China (43):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Hohhot
  - Research Site, Huzhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Quanzhou
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xining
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
  - Research Site, Zibo
  - Research Site, Zunyi
- Philippines (2):
  - Research Site, Iloilo City
  - Research Site, Quezon City
- South Korea (5):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Suwon

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D5180C00021-Primary CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00021&attachmentIdentifier=3f72a345-e246-4de4-8c5d-b0cf83127dc0&fileName=D5180C00021-Primary_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: D5180C00021-Final CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00021&attachmentIdentifier=2fd5959d-d1d1-4532-af2e-f258447dccb3&fileName=D5180C00021-Final_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: D5180C00021 SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00021&attachmentIdentifier=bdcb0f1d-99a8-47d7-8cca-967c2e36c7c1&fileName=D5180C00021_SAP_Redacted.pdf&versionIdentifier=
- See also: D5180C00021 CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00021&attachmentIdentifier=3ae5f974-d4c4-4d0c-949b-b0add12d16bb&fileName=D5180C00021_CSP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 401 participants were randomized at 74 sites in 3 Asian countries to receive treatment with tezepelumab 210mg Q4W or placebo.
Pre-assignment Details: Of the 401 randomized, 400 (99.8%) participants received treatment.
Groups:
- Tezepelumab 210mg Q4W: Tezepelumab administered every 4 weeks subcutaneously
- Placebo: Placebo administered subcutaneously
Period: Overall Study
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Started | 201 | 199
Completed | 186 | 168
Not Completed | 15 | 31
Not completed — Adverse Event | 1 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 8 | 21
Not completed — Due to COVID-19 pandemic | 5 | 2
Not completed — Protocol-specified withdrawal criterion met | 0 | 2
Not completed — Other than above | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tezepelumab 210mg Q4W | Placebo | Total
Number analyzed (Participants) | 201 | 199 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 166 | 167 | 333
  >=65 years | 35 | 32 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (12.4) | 54.3 (10.3) | 53.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 112 | 231
  Male | 82 | 87 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 201 | 199 | 400
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 201 | 199 | 400
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annual Asthma Exacerbation Rate (AERR)
Description: The annual exacerbation rate is based on exacerbations reported by the investigator in the eCRF over 52 weeks
Time Frame: Randomization to Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Events per year | 0.42 [0.30 to 0.59] | 1.63 [1.22 to 2.19]
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Negative Binomial Regression; Rate Ratio = 0.26, 95% CI 2-sided [0.17 to 0.39]

2. Secondary Outcome: Mean Change From Baseline in Pre-dose/Pre-bronchodilator (Pre-BD) Forced Expiratory Volume in 1 Second (FEV1) at Week 52
Description: Mean change from baseline in FEV1 as compared to placebo at Week 52. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Time Frame: Randomization to Week 52
Population: All participants from the Full Analysis Set with at least one change from baseline value at any post-baseline visit contributes to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 197
Litre | 0.35 (0.029) | 0.11 (0.030)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 0.24, 95% CI 2-sided [0.16 to 0.32]

3. Secondary Outcome: Mean Change From Baseline in Standardized Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(S)+12) Total Score at Week 52
Description: Mean change from baseline in AQLQ(S)+12 as compared to placebo at Week 52. The AQLQ(S)+12 is a questionnaire that measures the health-related quality of life experienced by asthma participants. The total score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. AQLQ(S)+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment).
Time Frame: Randomization to Week 52
Population: All participants from the Full Analysis Set with at least one change from baseline value at any post-baseline visit contribute to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 196
Scores on a scale | 1.29 (0.074) | 0.94 (0.076)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Least Squares Means Difference = 0.35, 95% CI 2-sided [0.14 to 0.55]

4. Secondary Outcome: Mean Change From Baseline in Asthma Control Questionnaire-6 (ACQ-6) Score at Week 52
Description: Mean change from baseline in ACQ-6 as compared to placebo at Week 52. The ACQ-6 captures asthma symptoms and short-acting β2-agonist use via subject-report. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses.
Time Frame: Randomization to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 196
Scores on a scale | -1.34 (0.058) | -1.03 (0.059)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Means Difference = -0.31, 95% CI 2-sided [-0.47 to -0.15]

5. Secondary Outcome: Mean Change From Baseline in Weekly Mean Daily Asthma Symptom Diary Score at Week 52
Description: Mean change from baseline in Asthma Symptom Diary score as compared to placebo at Week 52. The Asthma Symptom Diary comprises of 10 items (5 items in the morning; 5 items in the evening). Asthma symptoms during night time and daytime are recorded by the patient each morning and evening in the daily diary. A daily ASD score is the mean of the 10 items. A higher value indicates a worse outcome. Responses for all 10 items are required to calculate the daily ASD score; otherwise, it is treated as missing. For the 7-day average asthma symptom score, scoring is done with no imputation using the mean of at least 4 of the 7 daily ASD scores as a mean weekly item score. The 7-day average ASD score ranges from 0 to 4.
Time Frame: Randomization to Week 52
Population: All participants from the Full Analysis Set with at least one change from baseline value at any post-baseline week contribute to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Scores on a scale | -0.61 (0.036) | -0.44 (0.037)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Least Squares Means Difference = -0.16, 95% CI 2-sided [-0.27 to -0.06]

6. Secondary Outcome: Time to First Asthma Exacerbation
Description: Time to the first occurrence of asthma exacerbation post randomization, presented as number of participants with at least one asthma exacerbation reported in the eCRF
Time Frame: Randomization to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Participants | 45 | 89

7. Secondary Outcome: Mean Change From Baseline in Fractional Exhaled Nitric Oxide at Week 52
Description: Mean change from baseline in FENO (ppb) at week 52 to assess the effect of 210 mg of tezepelumab SC Q4W on biomarkers
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (Standard Error); unit: ppb
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 196
ppb | -15.88 (1.628) | -3.15 (1.658)

8. Secondary Outcome: Number of Participants With Asthma Specific Resource Utilization Over 52 Weeks
Description: Number of participants with asthma specific resource utilization (e.g. unscheduled physician visits, unscheduled phone calls to physicians, use of other asthma medications) over 52 weeks.
Time Frame: Randomization to Week 52
Measure: Number; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Participants
  Hospitalisation | 4 | 13
  Emergency room visit | 5 | 11
  Unscheduled visit to specialist | 36 | 75
  Home visit | 1 | 0
  Telephone call | 28 | 55
  Ambulance transport | 0 | 2

9. Secondary Outcome: Pharmacokinetics of Tezepelumab
Description: Mean serum trough PK concentrations taken pre-dose at each scheduled visit to evaluate the pharmacokinetics (PK) of tezepelumab
Time Frame: Baseline, Week 24, Week 52, Week 64
Population: PK Analysis Set: participants who received at least one dose of tezepelumab. The placebo arm is not applicable. Number analyzed at each timepoint is a subset of PK Analysis Set based on participants who had sample results available at that timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Tezepelumab 210mg Q4W
Number analyzed (Participants) | 198
ug/mL
  Baseline: number analyzed (Participants) | 196
  Baseline | 0 (0)
  Week 24: number analyzed (Participants) | 154
  Week 24 | 21.3513 (43.96)
  Week 52: number analyzed (Participants) | 144
  Week 52 | 21.2222 (41.51)
  Week 64: number analyzed (Participants) | 169
  Week 64 | 1.4450 (157.46)

10. Secondary Outcome: Mean Change From Baseline in EQ-5D-5L VAS Score at Week 52
Description: Mean change from baseline in EQ-5D-5L VAS at week 52. EQ-5D-5L visual analogue scale (VAS) allows participants to rate current health status on a scale of 0-100, with 0 being the worst imaginable health state.
Time Frame: At Week 52
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 196
Scores on a scale | 12.80 (1.009) | 9.67 (1.028)

11. Secondary Outcome: Mean Change From Baseline in Blood Eosinophils (Cells/uL) at Week 52
Description: Mean change from baseline in blood eosinophil counts at week 52 to assess the effect of 210 mg of tezepelumab SC Q4W on biomarkers.
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (Standard Error); unit: cells/uL
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 197
cells/uL | -193.44 (21.538) | -38.86 (21.984)

12. Secondary Outcome: Mean Change From Baseline in Total Serum IgE (IU/mL) at Week 52
Description: Mean change from baseline in IgE at week 52 to assess the effect of 210 mg of tezepelumab SC Q4W on biomarkers.
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (Standard Error); unit: IU/mL
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 200 | 197
IU/mL | -92.77 (27.460) | 0.30 (28.013)

13. Secondary Outcome: Mean Change From Baseline in Night Time Awakenings (Percentage) at Week 52
Description: Mean change from baseline in night time awakenings due to asthma at Week 52. Night time awakenings percentage is defined as number of nights with awakenings due to asthma and requiring rescue medication divided by number of nights with available data and multiplied by 100%. At least 4 out of 7 days of data is required to calculate a weekly mean.
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights with awakenings
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Percentage of nights with awakenings | -18.74 (1.035) | -15.99 (1.093)

14. Secondary Outcome: Immunogenicity of Tezepelumab
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline. Persistently positive is defined as positive at >=2 post baseline assessments (with >=16 weeks between the first and the last positive) or positive at last post baseline assessment. Transiently positive is defined as having at least one post baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Treatment boosted ADA defined as baseline positive ADA that was boosted to a 4 fold or higher level following treatment. Treatment emergent ADA defined as sum of treatment induced ADA and treatment boosted ADA.
Time Frame: Baseline to Week 64
Measure: Number; unit: Participants
Groups:
- Tezepelumab 210mg Q4W (China Cohort): Tezepelumab administered every 4 weeks subcutaneously; China cohort
- Placebo (China Cohort): Placebo administered subcutaneously; China cohort
- Tezepelumab 210mg Q4W (Non-China Cohort): Tezepelumab administered every 4 weeks subcutaneously; non-China cohort
- Placebo (Non-China Cohort): Placebo administered subcutaneously; non-China cohort
Arm/Group | Tezepelumab 210mg Q4W (China Cohort) | Placebo (China Cohort) | Tezepelumab 210mg Q4W (Non-China Cohort) | Placebo (Non-China Cohort)
Number analyzed (Participants) | 155 | 153 | 46 | 46
Participants
  ADA positive at baseline and/or post-baseline | 11 | 18 | 3 | 7
  Any baseline ADA positive | 10 | 14 | 2 | 5
  Only baseline ADA positive | 10 | 7 | 2 | 5
  Any post-baseline ADA positive | 1 | 11 | 1 | 2
  Both baseline and at least one post-baseline ADA positive | 0 | 7 | 0 | 0
  Treatment-induced ADA positive | 1 | 4 | 1 | 2
  Treatment-boosted ADA positive | 0 | 1 | 1 | 0
  TE-ADA positive | 1 | 5 | 1 | 2
  ADA persistently positive | 1 | 10 | 1 | 1
  ADA transiently positive | 0 | 1 | 0 | 1

15. Secondary Outcome: Mean Change From Baseline in Daily Rescue Medication Use (Weekly Means) at Week 52
Description: Daily rescue medication use is defined as: Number of night inhaler puffs + 2 x [number of night nebulizer times] + number of daytime inhaler puffs + 2 x [number of day nebulizer times]. Weekly means are calculated using at least 4 of 7 days of daily rescue medication use.
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (Standard Error); unit: Inhalations and nebulizers per week
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Inhalations and nebulizers per week | -0.81 (0.064) | -0.70 (0.066)

16. Secondary Outcome: Mean Change From Baseline in Home Based Morning Peak Expiratory Flow (PEF) at Week 52
Description: Mean change from baseline in home based morning PEF (L/min) at Week 52. Home PEF testing was performed by participant in the morning upon awakening and in the evening at bedtime using an electronic, hand-held spirometer. Weekly means are calculated using at least 4 of the 7 days of PEF data.
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
L/min | 46.70 (4.586) | 18.96 (4.730)

17. Secondary Outcome: Mean Change From Baseline in Home Based Evening Peak Expiratory Flow (PEF) at Week 52
Description: Mean change from baseline in home based evening PEF (L/min) at Week 52. Home PEF testing was performed by participant in the morning upon awakening and in the evening at bedtime using an electronic, hand-held spirometer. Weekly means are calculated using at least 4 of the 7 days of PEF data.
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 200 | 197
L/min | 42.14 (4.558) | 16.81 (4.700)

18. Secondary Outcome: Annual Asthma Exacerbation Rate Resulting in Emergency Room Visit or Hospitalization
Description: The annual exacerbation rate is based on exacerbations reported by the investigator that are associated with an emergency room visit, urgent care visit, or a hospitalization (where urgent care visit was captured as an emergency room visit on the eCRF).
Time Frame: Randomization to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Events per year | 0.07 [0.03 to 0.15] | 0.18 [0.09 to 0.34]

19. Secondary Outcome: Proportion of Participants Who Had no Asthma Exacerbations
Description: The proportion of participants who had no asthma exacerbations is presented as the percentage of participants with no exacerbations. This is defined as participants who meet both the following criteria: (1) completed the 52 week treatment period and (2) did not report an exacerbation during this period.
Time Frame: Randomization to Week 52
Measure: Number; unit: Percentage
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 201 | 199
Percentage | 74.6 | 50.3

ADVERSE EVENTS:
Time Frame: Adverse events is collected from time of signature of the informed consent form until end of study at Week 64.
Arm/Group | Tezepelumab 210mg Q4W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/201 | 2/199
Serious Adverse Events (participants affected / at risk) | 16/201 | 36/199
Other Adverse Events (participants affected / at risk) | 114/201 | 125/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab 210mg Q4W (N=201) | Placebo (N=199)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 4 (5)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 17 (27)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Myocardial bridging (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab 210mg Q4W (N=201) | Placebo (N=199)
Bronchitis (Infections and infestations) | 6 (6) | 7 (7)
Covid-19 (Infections and infestations) | 29 (30) | 25 (25)
Nasopharyngitis (Infections and infestations) | 11 (13) | 16 (26)
Pharyngitis (Infections and infestations) | 2 (2) | 7 (7)
Pneumonia (Infections and infestations) | 3 (3) | 9 (15)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 7 (7)
Respiratory tract infection (Infections and infestations) | 1 (1) | 8 (8)
Rhinitis (Infections and infestations) | 1 (1) | 6 (7)
Suspected covid-19 (Infections and infestations) | 16 (17) | 25 (25)
Upper respiratory tract infection (Infections and infestations) | 71 (127) | 68 (114)
Urinary tract infection (Infections and infestations) | 7 (11) | 7 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 9 (13)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7)
Gastritis (Gastrointestinal disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT03927157/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03927157/SAP_001.pdf